CLINICAL TRIAL: NCT04122209
Title: The Effect of Multiple Exercise Bouts During the Same Day (Continuous and High Intensity Intermittent Exercise), on Gastrointestinal Function, Appetite and Metabolic Response in Healthy Males: a Randomised Cross Over Trial
Brief Title: Does the Timing of When High Intensity Intermittent Exercise is Undertaken Matter?
Acronym: HIIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Lewis R Mattin, Postgraduate Teaching assistant (Nutritional Physiology), Manchester Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LRM-11619
Record Dates: First submitted 2019-09-03; First posted 2019-10-10 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Weight Loss; Weight Change, Body; Nutritional and Metabolic Disease
Keywords: Nutritional; Metabolic; Endocrine
MeSH Terms: conditions — Weight Loss; Body Weight Changes; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIE-First (Experimental): 60-min of exercise split into; firstly 30-min HIIE (10 x 1min of PPO, followed by 2-min rest). Secondly 30-min of continuous exercise (50% peak maximal oxygen uptake).
  Interventions: Other: HIIE-First
- Continuous-First (Experimental): 60-min of exercise split into; firstly 30-min of continuous exercise (50% peak maximal oxygen uptake). Secondly 30-min HIIE (10 x 1min of PPO, followed by 2-min rest)
  Interventions: Other: Continuous-First

INTERVENTIONS:
Other: HIIE-First — Multiple exercise bout during the same day; HIIE first followed by continuous exercise
  Arms: HIIE-First
Other: Continuous-First — Multiple exercise bout during the same day; Continuous exercise first followed by HIIE
  Arms: Continuous-First

SUMMARY:
The participants will visit the laboratory on 3 occasions, once for a preliminary visit and a further two occasions to complete experimental trials in a randomised order. The experimental trials will consist of cycling under two conditions; HIIE-First followed by Continuous (Trial-A) or Continuous-First followed by HIIE (Trial-B). Participants will be asked to standardise their diet for 24-hours and complete an overnight fast prior to visiting the laboratory. Participants will then complete 60-min of cycling split throughout the day into two 30-min bouts, HIIE or continuous cycling before breakfast followed by a 3.5 hour rest period before completing their remaining 30-min HIIE or Continuous cycling before lunch. Each experimental trail will last approximately 8 hours and begin at 08:00am. Throughout the trial measurements of subjective feelings of appetite, gastric emptying rate, substrate utilisation and regular blood samples will be taken. Post-trial nutritional and well-being questionnaires will be collected at 24-h post.

Study hypothesis

1. The order in which continuous and HIIE is undertaken will result in differences in gastric emptying rate after ingesting a semi-sold lunch?
2. Depending on which mode of exercise is undertaken first will result in different gastrointestinal hormone responses, metabolic responses and appetite responses throughout the trial day?
3. Will the order in which different modes of exercise, undertaken within the same day effect nutritional intake and well-being 24-h after both exercise bout have been completed?
4. Is substrate oxidation effected by the order in which multiple exercise bout of different modes are undertaken within the same day.

DETAILED DESCRIPTION:
There is a growing amount of literature committed to understanding if becoming more active will have beneficial effects on metabolic health; secondly do the traditional physical exercise and dietary approaches to managing obesity result in prolonged weight loss. The purpose of this study is to determine whether high intensity intermittent exercise (HIIE) and continuous exercise carried out in differing sequences within a day will have a beneficial health impact.

Participants will complete two 8h experimental trials in a randomised cross-over design. Each participant will complete 60-min of exercise in both trial arms; HIIE-First or Continuous-First separated by a minimum of 7 days. One trial will consist of a 30-min HIIE cycling session (10 x 1min of peak power output followed by 2min rest). After completion of this bout of exercise, participants will ingest a standardised breakfast. Following a rest period of 3h before completing the remaining 30-min of exercise (50% peak maximal oxygen uptake), before consuming a standardised semi-sold lunch meal. The second trial will be identical other than participates will undertake the continuous exercise first followed by the HIIE. Regular appetite, breath and blood samples will be taken throughout the trials. In The 24 hours following the end of each trial, participants will be asked to record their dietary intake and record their feeling of well-being documented on a questionnaire. There will be no long-term follow up following completion of the study.

Therefore, the aim of this research project is to identify whether the order of HIIE and continuous exercise separated within the day results in changes to gastrointestinal health, appetite, and metabolic responses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age between 18-40 years
3. Body mass index = <29.9 kg/m2
4. Non-smokers
5. No history of GI symptoms
6. Not consuming prescription medication, or no other relevant medical conditions assessed by a medical screening questionnaire.
7. Not vegan or lactose intolerant
8. Subsequently be physically active, in order to complete the trials.

Exclusion Criteria:

1. Not healthy
2. Female
3. Under 18 years
4. Over 40 years
5. Body mass index = >29.9 kg/m2;
6. Smokers
7. History of GI symptoms or disease,
8. Consuming prescription medication
9. Lactose Intolerant
10. Vegan
11. Subsequently not physically active, in order to complete the trials

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male participants will be recruited for this study, as we are unsure if hormonal responses between males and females would influence the outcomes within key measurements. Introducing females within this research area is important. However, for this current study we were particularly interested in data from male participates only
Enrollment: 12 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-05-18 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in gastric emptying rate over a 2-hour period | 9 breath samples will be collected at pre-Lunch (315 minutes), 345, 360, 375, 390, 405, 420, 435 and 450 minutes. Which is every 15 minutes for a two-hour period post-lunch.
  Gastric emptying rate of a semi-solid meal will be measured using the 13C breath test.
Changes in circulating levels of key gut hormones during the trial day | 10 samples will be collected at 0 (baseline), 30, 75, 135, 195, 255, 285, 315, 390, 450 minutes (End of trial)
  Hormones will be collected from serum blood samples
Changes in circulating levels of key metabolic markers during the trial day | 10 samples will be collected at 0 (baseline), 30, 75, 135, 195, 255, 285, 315, 390, 450 minutes (End of trial)
  Serum blood samples will be collected to measure Metabolic markers ( Glucose, triglycerides, Cholesterol and Non-esterified fatty acids)
Changes in substrate oxidation during the trial day | 8 measurements of substrate oxidation will be taken at 0 (baseline), 30, 135, 195, 255, 285, 390, and 450 minutes (End of trial)
  Substrate oxidation will be measured using a breath-by breath gas analyser for a 15-minutes period during each measurement
Changes in appetite using a visual analogue scales (VAS) questionnaire | 10 VAS questionnaires will be completed at 0 (baseline), 30, 75, 135, 195, 255, 285, 315, 390, 450 minutes (End of trial)
  Visual analogue scales will be used to measure subjective sensations of appetite. The VAS was composed of 6 questions asking: "how hungry do you feel?" "How full do you feel?" "How much do you think you can eat?" "How satisfied do you feel?" " How nauseous do you feel?" and " How bloated do you feel?". Horizontal lines 100 mm in length were anchored with "I am not hungry at all to I have never been more hungry," "Not at all full to totally full," "nothing at all to a lot," "I am completely empty to I can't eat another bite" " Not at all nauseous to Very nauseous" and " Not at all bloated to Very Bloated" at 0 mm and 100 mm, respectively.
Post trial energy intake | 24-hours post-trial total dietary intake
  24-hour post trial energy intake using weighed food intake dietary record

SECONDARY OUTCOMES:
Changes in well-being | 6 questionnaires will be completed; pre (0-minutes) and post first exercise bout (30-minutes), and pre (255-minutes) and post second exercise bout (285-minutes). End of the trial day (450-minutes), and 24-hours post-trial
  Well-being will be assessed with an in-house questionnaire. Before each trial session participants will answered the following questions: 1) how sore do your muscles feel ? 2) How fatigued do you feel today? 3) How is your mood? 4) How stressed do you feel today? 5) How sleepy do you feel?. Each question will be scored between 1 (low) and 7 (high). A sum of scores for the 5 questions will be used for data analysis.
Changes in perceived exertion | Perceived exertion will be asked 12 times; 6 during the first 30-minutes exercise period ( 5, 10, 15. 20, 25 and 30-minutes) and a further 6 times during the second exercise period (5, 10, 15, 20, 25 and 30-minutes
  Ratings of perceived exertion using the Borg scale will be recorded during exercise. Perceived exertion will be measured every 5-minutes during both 30-minutes exercise periods
Changes in heart rate during exercise | Continues exercise ( 5, 10, 15, 20, 25 and 30-minutes ) and Intermittent ( 1, 3, 6, 9, 12, 15, 18, 21, 24 and 27-minutes)
  Heart rate will be measured every 5-minutes during the continues exercise and every 3-minutes during the intermittent exercise

CONTACTS AND LOCATIONS:
Overall Officials: Gethin H Evans, PhD, Study Director — Manchester Metropolitan University
Locations (1):
- Manchester Metropolitan University, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Planned communication of results at a scientific conference. Planned publication in a high impact peer reviewed journal within 12 months of the completion of the study.IPD sharing statement: Participants level data is not expected to be available as this complies with the conditions of the ethical approval grated for this study

REFERENCES:
- [Background] Mattin LR, Yau AMW, McIver V, James LJ, Evans GH. The Effect of Exercise Intensity on Gastric Emptying Rate, Appetite and Gut Derived Hormone Responses after Consuming a Standardised Semi-Solid Meal in Healthy Males. Nutrients. 2018 Jun 19;10(6):787. doi: 10.3390/nu10060787. PMID 29921786
- [Background] McIver VJ, Mattin LR, Evans GH, Yau AMW. Diurnal influences of fasted and non-fasted brisk walking on gastric emptying rate, metabolic responses, and appetite in healthy males. Appetite. 2019 Dec 1;143:104411. doi: 10.1016/j.appet.2019.104411. Epub 2019 Aug 21. PMID 31445052
- [Background] McIver VJ, Mattin L, Evans GH, Yau AMW. The effect of brisk walking in the fasted versus fed state on metabolic responses, gastrointestinal function, and appetite in healthy men. Int J Obes (Lond). 2019 Sep;43(9):1691-1700. doi: 10.1038/s41366-018-0215-x. Epub 2018 Sep 24. PMID 30250241